CLINICAL TRIAL: NCT04775797
Title: A Double-Blind, Randomized, Placebo-Controlled, Single and Multiple Dose Study Evaluating the Safety, Tolerability, and Pharmacokinetics of AB-836, an HBV Capsid Inhibitor, in Healthy Subjects and Subjects With Chronic HBV Infection
Brief Title: Safety, Tolerability, and Pharmacokinetics of AB-836 in Healthy Subjects and Subjects With Chronic HBV Infection
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Safety
Sponsor: Arbutus Biopharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AB-836-001
Record Dates: First submitted 2021-02-24; First posted 2021-03-01 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Chronic Hepatitis
MeSH Terms: conditions — Hepatitis, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Single blind only (Participant) in Part 2b
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Part 1 (Healthy Subjects): Single Ascending Dose (SAD) (Experimental): Two cohorts (Cohorts A and B) of healthy subjects will receive single doses of AB-836/placebo in an alternating cohort design under fasted conditions. One additional treatment will be administered under fed conditions.
  Interventions: Drug: AB-836; Drug: Placebo
- Part 2a (Healthy Subjects): Multiple Ascending Dose (MAD) (Experimental): Participants in Cohorts C, D and E will receive a once daily dose of AB-836/placebo for 10 days
  Interventions: Drug: AB-836; Drug: Placebo
- Part 3 (Chronic Hepatitis B [CHB] Participants): MAD Cohorts F-H (Experimental): Participants in Cohorts F, G, and H will receive multiple doses of AB-836/placebo once daily for 28 days.
  Interventions: Drug: AB-836; Drug: Placebo
- Part 3 (Chronic Hepatitis B [CHB] Participants): MAD Cohort I (Experimental): Participants in Cohort I will receive multiple doses of AB-836/placebo once daily for 28 days in combination with ongoing nucleos(t)ide analog (NA) therapy.
  Interventions: Drug: AB-836; Drug: Placebo; Drug: Nucleos(t)ide Analogue
- Part 2b (Healthy Subjects): MAD (Experimental): Participants in Cohorts J will receive a once daily dose of AB-836/placebo for 35 days
  Interventions: Drug: AB-836; Drug: Placebo

INTERVENTIONS:
Drug: AB-836 — Capsules or Tablets
  Arms: Part 1 (Healthy Subjects): Single Ascending Dose (SAD)
Drug: Placebo — Capsules of Tablets
  Arms: Part 1 (Healthy Subjects): Single Ascending Dose (SAD)
Drug: AB-836 — Tablets
  Arms: Part 2a (Healthy Subjects): Multiple Ascending Dose (MAD); Part 2b (Healthy Subjects): MAD; Part 3 (Chronic Hepatitis B [CHB] Participants): MAD Cohort I; Part 3 (Chronic Hepatitis B [CHB] Participants): MAD Cohorts F-H
Drug: Placebo — Tablets
  Arms: Part 2a (Healthy Subjects): Multiple Ascending Dose (MAD); Part 2b (Healthy Subjects): MAD; Part 3 (Chronic Hepatitis B [CHB] Participants): MAD Cohort I; Part 3 (Chronic Hepatitis B [CHB] Participants): MAD Cohorts F-H
Drug: Nucleos(t)ide Analogue — Tablets
  Arms: Part 3 (Chronic Hepatitis B [CHB] Participants): MAD Cohort I

SUMMARY:
This three-part, Phase 1 protocol will be the first clinical study of AB-836. Parts 1 and 2a/b will be a Phase 1a SAD/MAD of AB-836 in healthy adult subjects. Part 3 will be a Phase 1b dose-ranging assessment of AB-836 in non-cirrhotic Chronic Hepatitis B (CHB) subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Subjects

  1. Male and Female (not of childbearing potential in Part 1 and 2a) subjects between 18 and 45 years old
  2. Free from clinically significant illness or disease as determined by their medical history, physical examination, vital signs, and clinical laboratory test results.
  3. BMI of 18-32 kg/m2.
* CHB Subjects:

  1. Male or female between 18 and 65 years old.
  2. Chronic HBV infection documented as a positive HBsAg, HBV DNA, or HBeAg test at least 6 months prior to the Screening Visit, or a historical liver biopsy consistent with chronic HBV infection
  3. For cohort F, G, H:

     1. HBV DNA ≥2,000 IU/mL at Screening (subjects may be either treatment-naïve or treatment-experienced but currently off-treatment).
     2. ALT ≤ 5x ULN
  4. For Cohort I:

     1. HBV DNA <LLOQ at Screening
     2. Subjects must have been receiving either TAF, TDF, or ETV consistently for ≥6 months prior to Day 1 and are willing to continue with the same NA treatment through the final study visit.
     3. ALT ≤ 2.5 x ULN
  5. HbsAg ≥250 IU/mL at screening

Exclusion Criteria:

* CHB Subjects

  1. Advanced fibrosis, cirrhosis or other signs of advanced liver disease as assessed by clinical history, ultrasound or FibroScan, or history of cirrhosis or any clinically significant medical condition associated with chronic liver disease.
  2. Co-infection with HIV or other non-B hepatitis viruses.
  3. Any clinically significant or unstable medical condition or illness that could confound study findings.
  4. Subjects who are unwilling to comply with protocol contraception requirements, and female subjects who are pregnant or breastfeeding.
  5. Previous treatment with a capsid inhibitor, core inhibitor, or core protein assembly modifier [CpAM or CAM]) within 6 months of the Day 1 visit, or prior treatment with an HBV-targeted siRNA or antisense oligonucleotide compound at any time.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2021-06-25 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2022-11-17 (Actual)

PRIMARY OUTCOMES:
Incidence of TEAEs | Up to 35 days after last dose of AB-836/placebo
Incidence of discontinuations due to AEs | Up to 35 days after last dose of AB-836/placebo
Incidence of lab abnormalities | Up to 35 days after last dose of AB-836/placebo

CONTACTS AND LOCATIONS:
Locations (15):
- Australia (2):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
- Canada (2):
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Toronto Liver Center, Toronto, Ontario
- Queen Mary Hospital, Hong Kong, Hong Kong
- Arensia Exploratory Medicine, Chisinau, Moldova
- New Zealand Clinical Research Auckland, Auckland, New Zealand
- South Korea (2):
  - Pusan National University Hospital, Busan
  - Asan Medical Center, Seoul
- Thailand (5):
  - Hospital For Tropical Diseases, Bangkok
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
  - Srinagarind Hospital, Khon Kaen
  - Naresuan University Hospital, Phitsanulok
- Medical Center of Limited Liability Company Arensia Exploratory Medicine, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: No